CLINICAL TRIAL: NCT05732103
Title: Phase 1/2 Multicenter, Open-Label Study of CTX-712 in Patients With Relapsed/Refractory Acute Myeloid Leukemia and Higher Risk Myelodysplastic Syndromes
Brief Title: A Study of CTX-712 in Relapsed/Refractory Acute Myeloid Leukemia and Higher Risk Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chordia Therapeutics, Inc. (Industry)
Collaborators: Theradex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C22-11236; CTX-712-CL-02 (Other: Chordia Therapeutics Inc.)
Record Dates: First submitted 2023-01-24; First posted 2023-02-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Cohort (Experimental): Drug: CTX-712 administered at 20 mg, 40 mg, 80 mg, 100 mg, 140 mg weekly, or 60 mg, 80 mg, 100 mg twice a week
  Interventions: Drug: CTX-712
- Initial Expansion Cohort (Experimental): Drug: CTX-712 administered at a dose to be determined from the data of dose escalation cohort
  Interventions: Drug: CTX-712
- Phase 2 (Experimental): CTX-712 administered at the recommended dose by the expansion cohort
  Interventions: Drug: CTX-712

INTERVENTIONS:
Drug: CTX-712 — CTX-712 will be provided as a 20 mg tablet for oral administration. Patients will take CTX-712 once or twice weekly, depending on their dose level assignment, during each 28-day cycle.

SUMMARY:
The goal of this phase 1/2 multicenter, open-label, single-arm dose escalation and expansion study is to assess the safety, tolerability, pharmacokinetic and pharmacodynamic profile of CTX-712 in patients with relapsed/refractory (R/R) acute myeloid leukemia (AML) and higher risk myelodysplastic syndromes (HR-MDS), or MDS/MPN (including CMML).

The phase 1 part of the study consists of sequential standard 3 + 3 dose escalation, where patients will receive ascending doses of CTX-712 to determine the recommended phase 2 dose (RP2D) for further clinical development. This is followed by initial expansion cohorts in AML and/or HR-MDS where patients will be treated with CTX-712 at the RP2D to gain further confidence in the selected dose level. Additional expansion cohorts may be initiated if considered necessary. After RP2D is determined, Drug-Drug-Interaction cohorts will be started.

The phase 2 part of the study will commence after the RP2D has been identified and confirmed and will evaluate therapeutic activity in R/R AML or R/R HR-MDS, in addition to confirmation of the safety profile.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years.
2. Diagnosis of AML, HR-MDS, or high marrow blast MDS/MPN (including CMML).
3. Prior treatment history must include 1-4 prior lines of therapy.
4. Adequate organ function evidenced by the following laboratory values:

   Creatinine clearance (CL) ≥60 mL/min Total serum bilirubin < 1.5 × upper limit of normal (ULN) Alanine aminotransferase (ALT) Aspartate aminotransferase(AST) < 2.5 × ULN White blood cell count at the time of the first dose <10 k/μL
5. Eastern Cooperative Oncology Group performance status ≤2.
6. Female patients of childbearing potential must have a negative pregnancy test within 7 days before study treatment initiation and if sexually active, agree to use a highly effective form of contraception throughout their participation during study treatment and up to 4 months after the last dose of study drug
7. Male patients with female partners of childbearing potential must, even if surgically sterilized, agree to practice effective barrier contraception during the entire study treatment period and through four months after the last dose of study drug, or practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant.

Exclusion criteria:

1. Diagnosis of acute promyelocytic leukemia.
2. Isolated extramedullary relapse (phase 2 only).
3. Active central nervous system (CNS) leukemia.
4. History of other malignancy.
5. Any of the following cardiopulmonary abnormalities:

   1. Myocardial infarction within six months prior to registration.
   2. New York Heart Association Class III or IV heart failure or known left ventricular ejection fraction < 50%.
   3. A history of familial long QT syndrome.
   4. Symptomatic atrial or ventricular arrhythmias not controlled by medications.
   5. QTcF ≥ 470 msec calculated according to institutional guidelines, unless due to underlying bundle branch block and/or pacemaker and with approval of the medical monitor.
   6. Known moderate to severe and clinically significant chronic obstructive pulmonary disease, interstitial lung disease and/or pulmonary fibrosis (e.g., requiring home oxygen therapy).
6. Pregnancy and/or lactation.
7. Major surgery (excluding placement of vascular access) within 4 weeks prior to first dose of CTX-712.
8. History of allogeneic organ transplantation (excluding cornea).
9. History of allogenic hematopoietic stem cell transplantation within 6 months of planned study treatment initiation and/or graft-versus host disease grade ≥ 1 following allogenic hematopoietic stem cell transplantation.
10. History of or chimeric antigen receptor T-cell therapy or other modified T cell therapy.
11. Active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus, hepatitis C virus, known human immunodeficiency virus, or acquired immunodeficiency syndrome related illness. Infections controlled with oral anti-infective agents, including prophylactic treatments, are allowed. Patient must be viral load negative.
12. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Frequency of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) related to CTX-712. | Adverse events are collected from time of informed consent through 28 days after last dose of CTX-712.
Phase 1: The maximum tolerated dose MTD. | Dose-limiting toxicities are collected during the first treatment cycle (28 days).
  MTD is the dose producing <33% of dose-limiting toxicities.
Phase 2: Complete remission rate, defined as the proportion of patients who achieve complete remission. | Measured from date of first dose to 28 days after last dose of CTX-712.

SECONDARY OUTCOMES:
Phase 1 and 2: Objective response rate, defined as the proportion of patients achieving a response. | Measured from date of first dose to 28 days after last dose of CTX-712.
  For AML: CR, CRi, PR, MLFS. For MDS: CR, PR, mCR, HI.
Phase 1 and 2: Duration of response. | Measure from documentation of tumor response to disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
Phase 1 and 2: Progression-free survival. | Measured from the date of initiating study treatment to the date of disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
Phase 1 and 2: Overall survival. | Measured from the date of initiating study treatment to the date of death from any cause, assessed up to 36 months.
Phase 1 and 2: Proportion of patients who transition to hematopoietic stem cell transplantation (HSCT). | Measured from the date of the last administration of CTX-712 until HSCT, or one year from the date of the start of administration of CTX-712.
Phase 1: Maximum observed plasma concentration (Cmax) of CTX-712. Plasma samples for PK analyses will be collected at predetermined time points and analyzed. | Pharmacokinetic evaluation performed in treatment Cycle 1 (cycle duration is 28 days).
Phase 1: Concentration before dose at steady state (Ctrough) of CTX-712. Plasma samples for PK analyses will be collected at predetermined time points and analyzed. | Pharmacokinetic evaluation performed in treatment Cycles 1, 2 and 4 (cycle duration is 28 days).
Phase 1: Area under the plasma concentration time curve (AUC) of CTX-712. Plasma samples for PK analyses will be collected at predetermined time points and analyzed. | Pharmacokinetic evaluation performed in treatment Cycle 1 (cycle duration is 28 days).
Phase 1: Volume of distribution (Vd) of CTX-712. Plasma samples for PK analyses will be collected at predetermined time points and analyzed. | Pharmacokinetic evaluation performed in treatment Cycle 1 (cycle duration is 28 days).
Phase 1: Elimination half-life of plasma concentration of CTX-712 at terminal phase (T1/2). Plasma samples for PK analyses will be collected at predetermined time points and analyzed. | Pharmacokinetic evaluation performed in treatment Cycle 1 (cycle duration is 28 days).
Phase 1: Clearance (CL) of CTX-712. Plasma samples for PK analyses will be collected at predetermined time points and analyzed. | Pharmacokinetic evaluation performed in treatment Cycle 1 (cycle duration is 28 days).
Phase 1: Measurement of the change in RNA splicing by CTX-712 in peripheral blood samples as pharmacodynamic markers. Peripheral blood samples for PD analyses will be collected at predetermined time points and analyzed. | Pharmacodynamic evaluation performed in treatment Cycle 1 (cycle duration is 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Comprehensive Cancer Center, Rochester, Minnesota
  - The University of Rochester, Rochester, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yokoyama H, Fukuhara N, Ando K, Iida H, Yamauchi T, Fukuhara S, Izutsu K, Tanoue Y, Yamamoto M, Tozaki H, Takahara E, Shoji S, Mizutani A, Morishita D, Oda RW, Miyake H, Yamamoto N. Phase I Study of Rogocekib in Patients with Relapsed or Refractory Hematologic Malignancies. Blood Adv. 2025 Oct 7:bloodadvances.2025017601. doi: 10.1182/bloodadvances.2025017601. Online ahead of print. PMID 41056522